CLINICAL TRIAL: NCT03212742
Title: Phase I/IIa Study of Concomitant Radiotherapy With Olaparib and Temozolomide in Unresectable High Grade Gliomas Patients
Acronym: OLA-TMZ-RTE-01
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OLA-TMZ-RTE-01
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Malignant Gliomas; Radiotherapy; PARP Inhibitor
MeSH Terms: conditions — Glioma | interventions — olaparib; Temozolomide; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMRT - Temozolomide - Olaparib (Experimental): The therapeutic regimen will be divided into 2 different periods:
  * Radiotherapy period The patient will start IMRT (60Gy/30fr/6 weeks), TMZ(Temozolomide) chemotherapy (75mg/m²/day), and olaparib on the same day, on a Monday (day 1), within 6 weeks after surgery. The daily dose of TMZ (75 mg/m²) will be continued until the end of radiotherapy (6 weeks) and olaparib will be continued with the same dose until 4 weeks after the end of IMRT, as a single agent.
  * Maintenance period TMZ will then be re-introduced 4 weeks after the end of IMRT at the dose of 150 mg/m2/day on days 1 to 5 every 28 days, for a total of 6 cycles. Concomitantly, olaparib will be daily given at the maintenance dose level up to confirmed disease progression or unacceptable toxicities.
  We propose 7 dose levels to reach the target dose of 400 mg per day (200 mg twice daily) of olaparib continuously
  Interventions: Drug: Olaparib; Drug: Temozolomide (TMZ); Radiation: IMRT (Intensity Modulated Radiation Therapy)

INTERVENTIONS:
Drug: Olaparib — We propose 7 dose levels to reach the target dose of 400 mg per day (200 mg twice daily) of olaparib continuously DL1 (starting dose level) : Olaparib 50 mg Q12H Monday to wednesday DL2 : Olaparib 100mg Q12H Monday to wednesday DL3: Olaparib 100mg Q12H Monday to friday DL4 : Olaparib 200mg Q12H Monday to wednesday DL5: Olaparib 200mg Q12H Monday to friday DL6: Olaparib 200mg Q12H, continously
Drug: Temozolomide (TMZ) — TMZ will be given at the dose of 75mg/m²/day during radiotherapy period. TMZ will be re-introduced 4 weeks after the end of radiotherapy at the dose of 150mg/m²/day on days 1 to 5 every 28 days, for a total of 6 cycles.
Radiation: IMRT (Intensity Modulated Radiation Therapy) — Radiotherapy consists of fractionated focal irradiation at a dose of 2 Gy per fraction given once daily five days per week over 6 weeks, for a total dose of 60 Gy by 3D- Intensity-Modulated RT (IMRT)

SUMMARY:
The Stupp protocol is the standard treatment of glioblastoma multiform (GBM) which prognosis remains poor.

The non-dividing nature of normal brain cells provides an opportunity to enhance the therapeutic ratio by combining radiation with inhibitors of replication-specific DNA repair pathways such poly(ADP-ribose) polymerase (PARP) inhibitors, thus inducing more cytotoxic effects of DNA-damage related to treatment modalities, including alkylating reagents like temozolomide (TMZ).

Olaparib, a potent PARP inhibitor, overcomes apoptotic resistance and sensitizes GBM cells for death receptor-mediated apoptosis induced by TRAIL (Tumor necrosis factor-Related Apoptosis Inducing Ligand). Moreover, inhibition of PARP activity increases cellular sensitivity to ionizing radiation: it was even suggested to be more pronounced in tumors than in normal tissue.

Lastly, progress in technical imaging and intensity-modulated-radiotherapy (IMRT) techniques provide new possibilities for sparing healthy tissues.

DETAILED DESCRIPTION:
HGGs are the most common and most aggressive primary brain tumor. There is a real need to improve care management of GBM patients. Attempts to achieve cure by increasing radiation dose result in unacceptable neurotoxicity. As for radiosensitizers, they can exacerbate normal tissue damage.

Since GBM represent a rapidly dividing cell population within the nonreplicating normal brain, the therapeutic ratio may be enhanced by specific radiosensitization of proliferating cells. Resistance to apoptosis is a paramount issue in the treatment of HGG. Targeting PARP by the inhibitors like olaparib can reduce proliferation and lowers the apoptotic threshold of HGG (effect showed in vivo and in vitro).

In this context, we propose a phase I-IIa trail to investigate the toxicity and efficacy of olaparib and TMZ concomitantly with radiotherapy in first line treatment of unresectable high risk HGG.

Correlation between treatment response and tumor profiling will allow us to identify biomarkers that can be useful in treatment improvement and/or present a prognostic value. Then, the transfer of this approach will be evaluated in terms of compatibility with the requirements of diagnostic.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent prior to any study specific procedures
* Histologically-confirmed diagnosis of glioblastoma (IDH-wildtype, IDH-mutant or NOS, except gliosarcoma), non resectable or partially resectable with a residual tumor on pre-radiotherapy MRI. The presence of a residual disease will be assessed by the radiologist on the pre-radiotherapy imaging as compared with initial imaging.
* IMRT must start within 6 weeks after histological diagnosis
* Age between 18 and 70 years ;
* Neurologically asymptomatic or pauci-symptomatic patients. Patients with moderated neurological symptoms without systemic corticosteroids treatment or with a stable dose of corticosteroids during the study as long as these were started at least 4 weeks prior to treatment can be included.
* Adequate bone marrow and organ function measured within 15 days prior to administration of study treatment as defined below:

  * Haemoglobin ≥ 10.0 g/dL with no blood transfusions (packed red blood cells and platelet transfusions) in the past 28 days before start of treatment
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L

    o No features suggestive of MDS/AML on peripheral blood smear
  * Platelet count ≥ 100 x 109/L
  * White blood cells (WBC) > 3x109/L
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal
  * Creatinine clearance estimated using the Cockcroft-Gault equation of ≥51 mL/min:

Estimated creatinine clearance = [(140-age(years)) x weight(kg) (x Fsex) ] / [serum creatinine (mg/dL) x 72] where Fsex=0.85 for females and Fsex=1 for males.

* ECOG performance status 0-2
* Patients must have a life expectancy ≥ 16 weeks.
* Women of childbearing potential (WOCBP) and men under efficient contraception during treatment and at least 6 months after the end of treatment.
* Evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1.
* Postmenopausal (if applicable) is defined as:

  * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments,
  * LH and FSH levels in the post-menopausal range for women under 50,
  * radiation-induced oophorectomy with last menses >1 year ago,
  * chemotherapy-induced menopause with >1 year interval since last menses,
  * or surgical sterilisation (bilateral oophorectomy or hysterectomy).
* Male patients and their partners, who are sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in, throughout the period of taking study treatment and for 3 months after last dose of study drug(s) to prevent pregnancy in a partner.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Subjects affiliated to an appropriate social security system

Exclusion Criteria:

* Any prior radiotherapy to brain
* Any prior chemotherapy or immunotherapy
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Candidate for a concomitant therapy with Tumor-Treating Fields during the maintenance treatment [70]
* Previous enrolment in the present study
* Participation in another clinical trial protocol within 30 days prior to enrolment;
* Any previous treatment with a PARP inhibitor, including olaparib.
* Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years
* Gadolinium hypersensitivity, or any contraindication to undergo MRI examination (Pacemaker, brain aneurysms clips)
* Patients who had no initial pre-surgery contrast enhanced MRI scan including the standard sequences (T1 non enhanced, T1 contrast enhanced, T2 FLAIR)
* Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 2 weeks from the last dose prior to study treatment. The patient can receive a stable dose of bisphosphonates for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment with study drug.
* Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
* Concomitant use of known strong (eg. phenobarbital, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, modafinil). The required washout period prior to starting olaparib is 5 weeks for phenobarbital and 3 weeks for other agents.
* Resting ECG with QTc > 470 msec detected on 2 or more time points within a 24 hour period or family history of long QT syndrome. If ECG demonstrates QTc > 470 msec, patient will be eligible only if repeat ECG demonstrates QTc ≤470 msec;
* Blood transfusions within 1 month prior to study start
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
* Major surgery within 14 days of starting study treatment and patients must have recovered from any effects of any major surgery.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression (untreated and unstable for at least 28 days prior to study entry), superior vena cava syndrome, extensive bilateral lung disease on HRCT scan or any psychiatric disorder that prohibits obtaining informed consent.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication (inflammatory bowel disease, major bowel resection …)
* Pregnant or breast feeding women.
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV) and are receiving antiviral therapy.
* Patients with known active hepatitis (i.e., Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids.
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
* For temozolomide treatment, patients with a known galactose intolerance, a Lapp lactase deficit or a glucose or galactose malabsorption syndrome (rare hereditary diseases)
* Patients with uncontrolled epileptic seizures.
* Neurological, addictive or psychiatric disorder;
* Lack of availability for clinical follow-up assessments;
* Persons protected by a legal regime (guardianship, trusteeship).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2017-09-04 (Actual); Primary Completion 2026-09-13 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The Recommended Phase II Dose (RP2D) - Phase I | The RP2D will be evaluated 4 weeks after the end of radiotherapy
  The primary objective for the phase I is to determine the Recommended Phase II Dose (RP2D) of olaparib combined with the Stupp protocol (TMZ and concomitant fractionated radiotherapy: 60Gy/30 fractions/6 weeks) in first line treatment of patients with unresectable high-grade gliomas
Overall survival - Phase II | 12 months after the first administration of treatment
  The primary objective for the phase II is to assess the 12-month overall survival of the combination

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - CHU, Amiens
  - Institut de Cancérologie de l'Ouest, Angers
  - CHU, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Guillaume le Conquérant, Le Havre
  - CH du Havre, Le Havre
  - GHBS, Lorient
  - Centre léon Bérard, Lyon
  - Hôpitaux universitaires La Pitié Salpétrière - Charles Foix, Paris
  - Institut Curie, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Institut Claudius Regaud, Toulouse

REFERENCES:
- [Background] Lesueur P, Lequesne J, Grellard JM, Dugue A, Coquan E, Brachet PE, Geffrelot J, Kao W, Emery E, Berro DH, Castera L, Goardon N, Lacroix J, Lange M, Capel A, Leconte A, Andre B, Leger A, Lelaidier A, Clarisse B, Stefan D. Phase I/IIa study of concomitant radiotherapy with olaparib and temozolomide in unresectable or partially resectable glioblastoma: OLA-TMZ-RTE-01 trial protocol. BMC Cancer. 2019 Mar 4;19(1):198. doi: 10.1186/s12885-019-5413-y. PMID 30832617
- [Result] Stefan D, Lesueur P, Lequesne J, Feuvret L, Bronnimann C, Castera M, Brachet PE, Hrab I, Ducloie M, Lacroix J, Lecornu M, Braux G, Christy F, Sunyach MP, Cohen-Jonathan Moyal E, Kao W, Faisant M, Emery E, Grellard JM, Sichel F, Laurent C, Fontanilles M, Clarisse B. Olaparib, Temozolomide, and Concomitant Radiotherapy for Partially Resected or Biopsy-Only Glioblastoma First-Line Treatment: Results from the OLA-TMZ-RTE-01 Phase I Study. Clin Cancer Res. 2025 Apr 1;31(7):1212-1222. doi: 10.1158/1078-0432.CCR-24-2974. PMID 39882966
- [Derived] Madhavan K, Balakrishnan I, Lakshmanachetty S, Pierce A, Sanford B, Fosmire S, Elajaili HB, Walker F, Wang D, Nozik ES, Mitra SS, Dahl NA, Vibhakar R, Venkataraman S. Venetoclax Cooperates with Ionizing Radiation to Attenuate Diffuse Midline Glioma Tumor Growth. Clin Cancer Res. 2022 Jun 1;28(11):2409-2424. doi: 10.1158/1078-0432.CCR-21-4002. PMID 35344040